CLINICAL TRIAL: NCT04225754
Title: Identification of Prognostic Parameters in Patients With " Senile " Amyloid Cardiomyopathy
Acronym: EVAMYLOSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.386; 2019-A03024-53 (Other: ID RCB)
Record Dates: First submitted 2019-12-30; First posted 2020-01-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aging of the population is a reality in our society, with a strong increase in the number of elderly patients hospitalized for heart failure in our institutions. Heart failure in these patients is more present than to younger patients, with preserved ejection fraction form (HFpEF). Aging is responsible for the onset of senile amyloid cardiomyopathy. This pathology is still imperfectly understood and its link with the increase in the frequency of HFpEF is important. In addition, specific treatments have just shown their effectiveness. It is therefore urgent to better identify the prognostic predictive parameters of this cardiomyopathy.

The pathophysiological involvement of the coronary microcirculation responsible for a true microvascular coronary disease (CMVD) has been described as predictive factor in all cardiomyopathies. However the implementation of preventive strategies and / or therapeutic of the coronary microcirculation dysfunction are limited because we lack of diagnostic tests available and applicable to large cohorts of patients.

Our team INSERM U1039 Radiopharmaceutiques Biocliniques in collaboration with the laboratory GIPSA-lab (Grenoble Images Speech Signal Automatique), laboratory specialized in the signal analysis, has developed a new method of analysis allowing to measure the coronary microcirculation dysfunction usable in SPECT thanks to the measurement of a myocardial perfusion heterogeneity index (IHPM) (patented technique). The 3C registry (NCT03479580) is a registry studying the prevalence and cardiovascular prognosis of macro and microcirculatory coronary artery disease using the latest coronary evaluation techniques in patient with cardiomyopathy. This registry deployed on interventional cardiology centers on the Alpine Arc is therefore also addressed to patients with senile cardiomyopathy. The data collected will provide a better understanding of the factors influencing the prognosis of senile cardiomyopathy and the prognostic contribution of the measurement of the IHPM will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, over 75 years old
* Social Security Affiliate
* Any patient with the diagnosis of cardiac amyloidosis after etiological evaluation in one of the 4 Alpin arc interventional cardiology centers (Grenoble University Hospital, GHM Grenoble, Annecy Hospital and Chambéry Hospital).
* Non opposition to participation

Exclusion Criteria:

* Concomitant ischemic cardiopathy with revascularization following cardiac scintigraphy exploration and subsequent coronary angiography.
* Concomitant non-amyloid non-ischemic cardiopathy (valvular cardiopathy)
* Major non-cardiac illness (eg, disseminated malignancy, severe neurological dysfunction at the time of diagnosis) or social condition that may preclude participation in a research study
* Major patient protected by law (article L1121-8)
* Person deprived of liberty (Article L1121-8)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient whose standardized etiological investigations have made the diagnosis of a senile amyloid cardiomyopathy in one of the 4 centers of interventional cardiology of the Alpine arc (CHU Grenoble, GHM Grenoble, CH Annecy, and CH Chambery)
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of myocardial perfusion heterogeneity index on mortality at 1 year in patients with senile cardiac amyloidosis. | 1 year
  Rate of occurrence of the primary endpoint: all-cause mortality at 1 year

SECONDARY OUTCOMES:
Prognostic value of IHMP on hospitalizations for heart failure in patients with senile cardiac amyloidosis. | 1 year
  Rate of secondary endpoint: hospitalization for heart failure
Prognostic value of IHPM on the quality of life in patients with senile cardiac amyloidosis | 1 year
  Minnesota Quality of Life Questionnaire
Relationships between IHPM and structural and functional measures in cardiac imaging in cardiac ultrasound | Inclusion
  Measurements in cardiac echography (longitudinal, radial and circumferential strain of the left ventricle in speckle tracking, left atrial strain in speckle tracking)
Relationships between IHPM and structural and functional measures in cardiac imaging in MRI. | Inclusion
  Measurement of IHPM in scintigraphy and measurements in cardiac MRI (right and left ventricular function, cardiac mass,% LV fibrosis).
Correlations between IHMP and geriatric frailty. | Inclusion
  grid SEGA-A (short emergency geriatric evaluation)
Relationships between IHPM in cardiac scintigraphy and the rhythmic evaluations. | inclusion
  Abnormality on holter frequency (atrial fibrillation and / or bradycardia requiring pacemaker implantation).
Comparison of IHPM between patients with amyloid senile cardiomyopathy and a control population paired with age and sex. | Inclusion
  Measurement of IHPM in myocardial scintigraphy in patients with senile cardiac amyloidosis and a control population paired with age and sex.
Side effect of tafamidis in this population | 1 year
  Rate of side effect in function of phenotype of patients (imaging, geriatric evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte CASSET, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided